CLINICAL TRIAL: NCT00540865
Title: Case Management and Problem Solving Therapy for Depressed, Homebound, Low-Income Elders
Brief Title: Effectiveness of Case Management Versus Case Management Plus Problem-solving Therapy to Treat Depression in Low-income Elders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH075897 (NIH); R01MH075897 (NIH); 0604008461 DATR A4-GPS; NCT00504868 (obsolete NCT alias)
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Depression
Keywords: Homebound Persons; Case Management; Problem Solving Therapy
MeSH Terms: conditions — Depression | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Participants will receive problem-solving therapy and case management
  Interventions: Behavioral: Problem-solving therapy (PST); Behavioral: Case management (CM)
- B (Active Comparator): Participants will receive case management
  Interventions: Behavioral: Case management (CM)

INTERVENTIONS:
Behavioral: Problem-solving therapy (PST) — The premise of PST is that psychotherapies implicitly help people to become better managers of their lives, in effect, to become better at solving problems. Unlike Case Management (CM) that seeks to increase its clients' availability and utilization of resources, PST focuses on the patients themselves and helps them develop skills in identifying, prioritizing, and solving problems, and thereby creates a sense of empowerment. Although CM and PST have different theoretical premises, they both focus on the resolution of concrete problems promoting depression.
  Arms: A
Behavioral: Case management (CM) — Different types of CM exist, but all share the theme of helping individuals cope with their illnesses through linkage to social services, advocacy, rehabilitation, and ongoing support during recovery from illnesses. CM will consist of the following components: 1) socialization to treatment; 2) needs assessment; 3) psychoeducation about depression; 4) service planning; 5) linkage to social services; 6) help with access to health care; 7) advocacy; and 8) exploration of barriers that perpetuate unmet needs.

SUMMARY:
This study will compare the effectiveness of case management combined with problem-solving therapy (CM-PST) versus case management (CM) alone for assisting elderly people with depression.

DETAILED DESCRIPTION:
Depression is a common mental disorder that affects many low-income elders. Many elders suffer from multiple chronic illnesses and often must deal with social and financial hardships as they continue to age. Rates of diagnosis and treatment for depression within the elderly population are low. This may be because elders are embarrassed to discuss their symptoms with their doctor and assume sadness and anxiety are a normal part of the aging process. However, depression is not a normal consequence of aging. Furthermore, it can severely impact people's lives, sleep patterns, concentration, and energy levels. This study will compare the effectiveness of case management combined with problem-solving therapy (CM-PST) versus case management (CM) alone for assisting elderly people diagnosed with depression.

CM involves identifying a person's particular needs and working with a case worker to plan and implement specific resources and services that will meet those needs. PST emphasizes the social context of an individual's situation through problem-solving and behavior change techniques. Recent studies have suggested that combining CM with PST may have a mutually beneficial effect on depressed, low-income elders. CM can help elders with their social and financial needs, and PST can improve their ability to cope with stressful events and utilize their new resources.

Participants in this open-label study will be randomly assigned to receive 12 sessions of either CM or CM-PST. Both treatments will be delivered at the participant's home by a trained case worker. Participants assigned to receive CM will focus on increasing their resources and reducing adversity. The case worker will help participants determine the causes of their unmet needs, create an action plan to meet those needs, encourage the use of services, and possibly advise their family members and health care providers to help facilitate the use of those services. Participants assigned to CM-PST will undergo a needs assessment during the first session to develop a problem-solving plan that will be implemented over the next 11 sessions. Each session will include instruction on how to use the PST approach to solve problems identified by both the therapist and participant. All participants will undergo a neuropsychological exam and complete psychological and physical functioning questionnaires prior to treatment and at Weeks 3, 6, 12, and 24.

ELIGIBILITY:
Inclusion Criteria:

* Receives home-delivered meal service
* Has at least one instrumental activity of daily living (IADL) impairment
* Meets Diagnostic and Statistical Manual of Mental Disorders (DSM)IV criteria for unipolar major depression
* Considered low income (30% of the local median income)
* Has a need for social services
* Experiences problem-solving difficulties
* Speaks English

Exclusion Criteria:

* Diagnosis of psychotic depression or experiences delusions
* Suicidal
* Diagnosed with any Axis I psychiatric disorder other than unipolar major depression
* History of substance abuse
* Axis II diagnosis of antisocial personality
* History of psychiatric disorders other than unipolar major depression or generalized anxiety disorder, such as bipolar disorder, hypomania, or dysthymia
* Diagnosed with dementia
* Acute or severe medical illness, such as delirium, metastatic cancer, major surgery, stroke, heart attack, or decompensated heart, liver, or kidney failure within 3 months of study entry
* Use of drugs known to cause depression, such as steroids, reserpine, alpha-methyl-dopa, tamoxifen, or vincristine
* Use of antidepressants
* Currently receiving psychotherapy
* Inability to perform any of the activities of daily living (ADLs) even with assistance
* Aphasia interfering with communication

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2007-05; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Depression | Measured at pretreatment and Weeks 3, 6, 9, 12, and 24

SECONDARY OUTCOMES:
Disability | Measured at pretreatment and Weeks 3, 6, 9, 12, and 24

CONTACTS AND LOCATIONS:
Overall Officials: George S. Alexopoulos, MD, Principal Investigator — Weill Medical College of Cornell University; Patricia A. Arean, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California - San Francisco, San Francisco, California
  - Weill Medical College of Cornell University, White Plains, New York

REFERENCES:
- [Derived] Solomonov N, Kerchner D, Bein O, Lee CE, Diaz JL, Ciarleglio A, Kim S, Sirey JA, Gunning FM, Raue PJ, Banerjee S, Arean PA, Alexopoulos GS. Precision Assignment to Psychosocial Interventions for Late-Life Depression: An Automated Treatment Decision Rule. JAMA Psychiatry. 2025 Nov 1;82(11):1075-1084. doi: 10.1001/jamapsychiatry.2025.2518. PMID 40960814
- [Derived] Arean PA, Hallgren KA, Jordan JT, Gazzaley A, Atkins DC, Heagerty PJ, Anguera JA. The Use and Effectiveness of Mobile Apps for Depression: Results From a Fully Remote Clinical Trial. J Med Internet Res. 2016 Dec 20;18(12):e330. doi: 10.2196/jmir.6482. PMID 27998876
- [Derived] Anguera JA, Jordan JT, Castaneda D, Gazzaley A, Arean PA. Conducting a fully mobile and randomised clinical trial for depression: access, engagement and expense. BMJ Innov. 2016 Jan;2(1):14-21. doi: 10.1136/bmjinnov-2015-000098. PMID 27019745
- [Derived] Arean PA, Raue PJ, McCulloch C, Kanellopoulos D, Seirup JK, Banerjee S, Kiosses DN, Dwyer E, Alexopoulos GS. Effects of Problem-Solving Therapy and Clinical Case Management on Disability in Low-Income Older Adults. Am J Geriatr Psychiatry. 2015 Dec;23(12):1307-1314. doi: 10.1016/j.jagp.2015.04.005. Epub 2015 Apr 24. PMID 26628206
- [Derived] Alexopoulos GS, Raue PJ, McCulloch C, Kanellopoulos D, Seirup JK, Sirey JA, Banerjee S, Kiosses DN, Arean PA. Clinical Case Management versus Case Management with Problem-Solving Therapy in Low-Income, Disabled Elders with Major Depression: A Randomized Clinical Trial. Am J Geriatr Psychiatry. 2016 Jan;24(1):50-59. doi: 10.1016/j.jagp.2015.02.007. Epub 2015 Feb 17. PMID 25794636